CLINICAL TRIAL: NCT04609332
Title: Association of Endothelial Damage and Angiogenesis Biomarkers With Morbidity and Mortality in SARS-CoV-2 Infection
Brief Title: Endothelial Damage and Angiogenesis Biomarkers During COVID-19
Status: Completed | Type: Observational
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Felipe Andrés Maldonado Caniulao, Principal Investigator, University of Chile
Other Study IDs: OAIC 1164/20
Record Dates: First submitted 2020-10-23; First posted 2020-10-30 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Covid19; Angiogenesis; Endothelial Dysfunction; Cardiovascular Morbidity
Keywords: Syndecan-1; Thrombomodulin; VEFG; ANG-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Endothelial damage and angiogenic biomarkers — Blood samples for biomarkers study

SUMMARY:
Severe SARS-CoV-2 disease is characterized by a progressive hypoxemic respiratory failure. Autopsies from these patients show severe endothelial damage with extensive vascular thrombosis, microangiopathy, and occlusion of alveolar capillaries and, finally, evidence of new vessel growth through intussusceptive angiogenesis.

This research aims to study endothelial damage and angiogenesis biomarkers and its association with major cardiovascular events.

DETAILED DESCRIPTION:
To study the presence of endothelial damage and angiogenic biomarkers with major cardiovascular events, the investigators will perform an observational study to evaluate plasma biomarkers concentrations in Covid-19 patients hospitalized in critical care units.

After ethical review board approval, the investigators will select 40 patients admitted to intensive care units (ICU). After patient written consent or if the participants are unable to consent, after a relative subrogated acceptance, the investigators will collect blood samples in the first 24 hrs and on the 10th day of hospitalization.

Venous blood samples are collected. After obtaining all samples, serum Syndecan-1, thrombomodulin, ANG-2, FGF basic, HGF, IL-8, PDGF-BB, TIMP-1, TIMP-2, TNFα y VEGF will be determined by a researcher blinded to the patient using commercially available Elisa kits. The concentration of each biomarker at each sample time will be compared. The investigators will observe clinical outcomes after one, 3, 6, and 12 months after the hospitalization.

The investigators found no previous data of this measurement in the COVID-19 scenario. In this observational study, the investigators select a sample size on convenience for the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years
2. Patient with a diagnosis of COVID-19 confirmed by PCR
3. Patient with radiological image suggestive of COVID-19 with pending confirmation
4. Need for ventilatory support with oxygen therapy by HFNC (High-flow nasal cannula)
5. Need for invasive mechanical ventilation.

Exclusion Criteria:

1. Patient with an image suggestive of COVID-19 with negative PCR
2. Anticoagulation users before admission for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will include Covid 19 patients admitted to ICU with the need for oxygen and ventilatory support. Blood plasma biomarkers will be obtained on the first and 10th day of hospitalization. Information on major cardiac events will be obtained from the patient clinical file and by phone interview after hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-09-26 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Syndecan-1 concentration at 10th day | 24 Hours, 10 Days
  Elevation of plasma Syndecan-1

SECONDARY OUTCOMES:
Change from Baseline ANG-2 concentration at 10th day | 24 Hours, 10 Days
  Elevation of plasma ANG-2
Change from Baseline FGF basic concentration at 10th day | 24 Hours, 10 Days
  Elevation of plasma FGF basic
Change from Baseline HGF concentration at 10th day | 24 Hours, 10 Days
  Elevation of plasma HGF
Change from Baseline IL-8 concentration at 10th day | 24 Hours, 10 Days
  Elevation of plasma IL-8
Change from Baseline PDGF-BB concentration at 10th day | 24 Hours, 10 Days
  Elevation of plasma PDGF-BB
Change from Baseline TIMP-1 concentration at 10th day | 24 Hours, 10 Days
  Elevation of plasma TIMP-1
Change from Baseline TIMP-2 concentration at 10th day | 24 Hours, 10 Days
  Elevation of plasma TIMP-2
Change from Baseline TNFα concentration at 10th day | 24 Hours, 10 Days
  Elevation of plasma TNFα
Change from Baseline VEGF concentration at 10th day | 24 Hours, 10 Days
  Elevation of plasma VEGF
Change from Baseline Thrombomodulin concentration at 10th day | 24 Hours, 10 Days
  Elevation of plasma Thrombomodulin
Major cardiovascular events | 1 month, 3 months, 6 months 12 months.
  Acute coronary syndrome, myocardial injury, pulmonary embolism, and death.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Maldonado, M.D., M.Sc., Principal Investigator — Hospital Clínico de la Universidad de Chile
Locations (1):
- Hospital Clínico de la Universidad de Chile, Independencia, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maldonado F, Morales D, Diaz-Papapietro C, Valdes C, Fernandez C, Valls N, Lazo M, Espinoza C, Gonzalez R, Gutierrez R, Jara A, Romero C, Cerda O, Caceres M. Relationship Between Endothelial and Angiogenesis Biomarkers Envisage Mortality in a Prospective Cohort of COVID-19 Patients Requiring Respiratory Support. Front Med (Lausanne). 2022 Mar 16;9:826218. doi: 10.3389/fmed.2022.826218. eCollection 2022. PMID 35372407